CLINICAL TRIAL: NCT06361290
Title: Diaphyseal Reconstruction Techniques of Lower Limbs in Childhood Malignant Tumors - Induced Membrane Technique Versus Vascularized Fibula Grafts
Brief Title: Diaphyseal Reconstruction of Malignant Tumors in Children
Acronym: RDTM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231703
Record Dates: First submitted 2024-03-28; First posted 2024-04-11 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-04

CONDITIONS: Childhood Malignant Tumors of Lower Limbs
Keywords: Diaphyseal reconstruction techniques; Induced membrane technique; Vascularized fibula; Vascularized fibula grafts; Malignant tumors; Childhood
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients under 18 years of age treated between 1986 and 2017 for malignant bone tumors of the lower limb (femur or tibia), diaphyseal or metaphyseal-diaphyseal and having benefited from diaphyseal resection of the tumor with biological reconstruction by either Membrane Induced, Fibula Vascularized and or Vascularized Fibula associated with an Allograft and having had a minimum follow-up of 5 years.
  Interventions: Other: Data collection from hospital medical records

INTERVENTIONS:
Other: Data collection from hospital medical records — Data collection from hospital medical records of patients concerning the 5 years following the resection of the tumor.

SUMMARY:
Primary malignant bone tumors represent 5% of malignant tumors in children, 90% of which are osteosarcomas or Ewing sarcomas.

The objective of oncological resection is local control of the disease. Excision of the entire tumor should make it possible to maintain good function of the limb, minimizing morbidity, and promoting acceptance by the patient.

Biological reconstructions offer the best long-term functional results. Several possibilities are then available: the Induced Membrane technique, the Vascularized Fibula and Vascularized Fibula associated with an Allograft.

Until today, no reconstruction technique in children has proven its superiority over another and no decision-making algorithm for therapeutic care has been determined based on the importance of the bone resection and the affected segment in diaphyseal tumor reconstruction surgery of the lower limb.

The aim of the present research is to compare the three techniques concerning the consolidation aspect, the reoperation rates, the rates of bone complications, septic, and the functional results by the study of the medical files of approximately 90 patients operated between 1986 and 2017.

DETAILED DESCRIPTION:
Primary malignant bone tumors represent 5% of malignant tumors in children, 90% of which are osteosarcomas or Ewing sarcomas.

The diagnosis of a bone tumor is based on the clinical, radiological and biopsy comparison.

The main issue in the treatment of malignant tumors is the vital prognosis and secondarily the functional prognosis. Historically, primary malignant bone tumors have been treated by amputation.

The tumor resection, thanks to advances in chemotherapy since the 1970s, today shows survival rates identical to radical techniques. The goal of surgery is local control of the disease. The excision of the entire tumor should make it possible to maintain good function of the limb, in particular to minimize morbidity, and promote acceptance by the patient. Biological reconstructions offer the best long-term functional results. Several possibilities are then available: the Induced Membrane, the Vascularized Fibula and the Vascularized Fibula associated with an Allograft.

Until today, no reconstruction technique in children has proven its superiority over another and no decision-making algorithm for therapeutic care has been determined based on the importance of the bone resection and the affected segment in diaphyseal tumor reconstruction surgery of the lower limb.

The aim of the study is to compare the 3 diaphyseal reconstruction techniques in the context of malignant tumors in children, and to fill this gap, by providing a decision tree allowing this choice to be made. The comparison concerns the consolidation aspect, the reoperation rates, the rates of bone complications, septic, and the functional results by the study of the medical files of approximately 90 patients operated between 1986 and 2017. The hypothesis of the study is that one of the techniques offers better consolidation rates in major resections, and that adjuvant oncological treatments modify the results that can be expected from these different techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 years old with a malignant bone tumor of the lower limb (femur or tibia), diaphyseal or metaphyseal-diaphyseal
* Patients operated between 1986 and 2017 for a diaphyseal resection of the tumor with biological reconstruction using either Induced Membrane, Vascularized Fibula and Vascularized Fibula associated with an Allograft
* Patient with a minimum follow-up of 5 years

Exclusion Criteria:

* Patient who died within 5 years or who had a follow-up of less than 5 years following the reconstruction procedure
* Patient with joint damage
* Patient over 18 years old at the time of surgery
* Patient who had an isolated reconstruction of the fibula
* Opposition of adult patients/holders of parental authority of minor patients to whom the study information note was sent, to the use of the patient's medical data for the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Historical cohort of all patients treated for a malignant bone tumor of the lower limb between 1986 and 2017 in the AP-HP Necker-Enfants Malades or Armand Trousseau hospitals, part of the oncological follow-up of which was possibly carried out at the Institut Gustave Roussy or the Institut Curie.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Duration of bone consolidation period | 5 years
  Radiological consolidation times based on follow-up radiographs will be compared to the size of the bone resections in order to establish the healing index. The deadlines for providing support to members will also be collected.

SECONDARY OUTCOMES:
Rate of surgical re-intervention | 5 years
  The rates of septic, transfusional and immediate intraoperative complications of each surgery will be compared. The recovery rate for sepsis will also be considered. Neurological and vascular complications will also be compared. The total number of interventions will be counted.
Short- and long-term complication rates | 5 years
  Bone complications will be noted: fractures, pseudarthrosis, axial deviation and stress fractures will be noted and compared between the techniques. Secondary axial deviation and lower limb length inequalities will also be the subject of a comparative study in long-term follow-up.
  Other rates of septic or other complications will also be noted.
Long-term functional results | 5 years
  Long-term functional results will be described: joint range of motion is measured clinically at the hip, knee and ankle and reported in degrees from standardized anatomical positions, a VAS assessment of pain is performed, length inequality is measured radiologically and reported in millimeters on based on the non-operated limb, an MSTS score is performed (Musculoskeletal Tumor Society Rating Scale), an Enneking score is also performed.
Relationship between radiotherapy and biological reconstruction result | 5 years
  To demonstrate the effect of adjuvant oncological treatments, the type of tumor and adjuvant and neoadjuvant treatment will be taken into account. In particular the presence or absence of post-operative radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Haumont, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Eric Mascard, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Armand-Trousseau, Paris
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stiller CA, Bielack SS, Jundt G, Steliarova-Foucher E. Bone tumours in European children and adolescents, 1978-1997. Report from the Automated Childhood Cancer Information System project. Eur J Cancer. 2006 Sep;42(13):2124-35. doi: 10.1016/j.ejca.2006.05.015. PMID 16919776
- [Background] Arndt CA, Crist WM. Common musculoskeletal tumors of childhood and adolescence. N Engl J Med. 1999 Jul 29;341(5):342-52. doi: 10.1056/NEJM199907293410507. No abstract available. PMID 10423470
- [Background] Hameed M, Dorfman H. Primary malignant bone tumors--recent developments. Semin Diagn Pathol. 2011 Feb;28(1):86-101. doi: 10.1053/j.semdp.2011.02.002. PMID 21675380
- [Background] Whelan JS, Jinks RC, McTiernan A, Sydes MR, Hook JM, Trani L, Uscinska B, Bramwell V, Lewis IJ, Nooij MA, van Glabbeke M, Grimer RJ, Hogendoorn PC, Taminiau AH, Gelderblom H. Survival from high-grade localised extremity osteosarcoma: combined results and prognostic factors from three European Osteosarcoma Intergroup randomised controlled trials. Ann Oncol. 2012 Jun;23(6):1607-16. doi: 10.1093/annonc/mdr491. Epub 2011 Oct 19. PMID 22015453
- [Background] Le Nen D, Dubrana F, Hu W, Prud'homme M, Lefè;vre C. Fibula vascularisée. Techniques, indications en orthopédie et traumatologie. EMC - Tech Chir - Orthopédie - Traumatol. 2006;1(1):1-10.
- [Background] Hariri A, Mascard E, Atlan F, Germain MA, Heming N, Dubousset JF, Wicart P. Free vascularised fibular graft for reconstruction of defects of the lower limb after resection of tumour. J Bone Joint Surg Br. 2010 Nov;92(11):1574-9. doi: 10.1302/0301-620X.92B11.23832. PMID 21037355